CLINICAL TRIAL: NCT06261684
Title: Intralesional Acyclovir Versus Cryotherapy in the Treatment of Plantar Warts. A Randomized Controlled Trial.
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Basant Ahmed Mohamed Abdelaal Helal, Dermatology Resident, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-259-2023
Record Dates: First submitted 2023-10-06; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Plantar Wart
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intralesional Acyclovir (Experimental): Intralesional acyclovir will be prepared by diluting 1 ampoule of Acyclovir 250mg into 3.5ml of saline solution to achieve a concentration of approximately 70mg/ml. Then 0.1ml will be injected intra-lesionally into the base of the wart. Any hyperkeratotic lesions should be pared before the treatment. This process will be repeated every 2 weeks for 5 sessions, and can be discontinued if complete resolution is achieved early.
  Interventions: Drug: Intralesional Acyclovir
- Cryotherapy (Active Comparator): Patients allocated to Group B will undergo cryotherapy using a liquid nitrogen spray gun. Any hyperkeratotic lesions should be pared before the treatment. Two freeze-thaw cycles will be applied each session, the spray gun should be held 1cm away from the wart and maintained until the wart and the 1-3mm of surrounding skin shows freezing, and each cycle should last 15 seconds. Next, the lesion will be left to thaw completely before starting the second cycle. This process will be repeated every 2 weeks for 5 sessions, and can be discontinued if complete resolution is achieved early
  Interventions: Device: Cryotherapy

INTERVENTIONS:
Drug: Intralesional Acyclovir — Intralesional Acyclovir in plantar warts
  Arms: Intralesional Acyclovir
Device: Cryotherapy — Cryotherapy of plantar warts
  Arms: Cryotherapy

SUMMARY:
The goal of this prospective randomized controlled study is to study the safety and efficacy of intralesional acyclovir compared to cryotherapy in plantar warts. The main questions needed to be answered are:

1. Is Intralesional acyclovir safe for plantar warts?
2. Is Intralesional acyclovir more efficient in treating plantar warts compared to cryotherapy?

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older, of both genders, with plantar warts

Exclusion Criteria:

* Patients on systemic treatment for warts eg. Acitretin, Acyclovir
* Hypersensitivity to Acyclovir
* Previous treatment to the same wart during the last 3 months
* Immunocompromised patients (as HIV, steroid intake, uncontrolled diabetes, etc.)
* Pregnant and breastfeeding females
* Cognitively impaired patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Cure rate | 10 weeks (5 sessions max)
  Number of patients healed after completion of the sessions
Recurrence rate | 24 weeks
  Number of patients had recurred plantar warts after receiving the treatment
Patient satisfaction score | 10 weeks
  Patient satisfaction questionnaire score

SECONDARY OUTCOMES:
Correlation of treatment with number of ipsilateral warts | 10 weeks
  Number of warts increased, decreased or stationary
Correlation of treatment with age | 10 weeks
  Percentage of patients successfully treated in each age group (Young 18-32 years; Middle age 33-46, Old age 47-60
Correlation of treatment with gender | 10 weeks
  Percentage of successfully treated male to female patients
Correlation of treatment with size of the wart | 10 weeks
  Percentage of successful treatment compared to the size of the wart

CONTACTS AND LOCATIONS:
Overall Officials: Shahira Ramadan, Professor, Study Chair — Cairo University; Yousra Azzazi, Lecturer, Study Director — Cairo University
Locations (1):
- Cairo University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elsayed A, Nassar A, Marei A, Hoseiny HAM, Alakad R. Intralesional Acyclovir: A Potential Therapeutic Option for Cutaneous Warts. J Cutan Med Surg. 2022 Jan-Feb;26(1):25-30. doi: 10.1177/12034754211037998. Epub 2021 Aug 19. PMID 34412535
- [Background] Garcia-Oreja S, Alvaro-Afonso FJ, Tardaguila-Garcia A, Lopez-Moral M, Garcia-Madrid M, Lazaro-Martinez JL. Efficacy of cryotherapy for plantar warts: A systematic review and meta-analysis. Dermatol Ther. 2022 Jun;35(6):e15480. doi: 10.1111/dth.15480. Epub 2022 Apr 6. PMID 35365922